CLINICAL TRIAL: NCT04078074
Title: Occlusal Stabilization Splints and Sleep Disordered Breathing
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of funds
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Aaron Glick, Clinical Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-DB-19-0444
Record Dates: First submitted 2019-09-01; First posted 2019-09-04 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Sleep Bruxism
MeSH Terms: conditions — Sleep Bruxism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (3):
- Maxillary OSS (Experimental)
  Interventions: Device: Maxillary OSS
- Mandibular OSS (Experimental)
  Interventions: Device: Mandibular OSS
- Modified farrar splint (Experimental)
  Interventions: Device: Modified farrar splint

INTERVENTIONS:
Device: Maxillary OSS — Maxillary OSS will be a night guard for the top teeth. Digital impressions will be taken at the first appointment. After delivery appointment the patient will take home a sleep test monitor and bruxism monitor to record respiration and muscle activity during sleep.This will be a 2 night sleep study (Night A will be without splint and Night B will be with splint). Therefore, the patient will sleep with the mouth guard one night and the monitoring device two nights. Subjects will also undergo cone beam computed tomography (CBCT) airway imaging with and without splint.
  Arms: Maxillary OSS
Device: Mandibular OSS — Mandibular OSS will be a night guard for the bottom teeth.Digital impressions will be taken at the first appointment. After delivery appointment the patient will take home a sleep test monitor and bruxism monitor to record respiration and muscle activity during sleep.This will be a 2 night sleep study (Night A will be without splint and Night B will be with splint). Therefore, the patient will sleep with the mouth guard one night and the monitoring device two nights. Subjects will also undergo CBCT airway imaging with and without splint.
  Arms: Mandibular OSS
Device: Modified farrar splint — Modified farrar splint will be a night guard for the top teeth that positions and maintains the lower jaw in a more forward position.Digital impressions will be taken at the first appointment. After delivery appointment the patient will take home a sleep test monitor and bruxism monitor to record respiration and muscle activity during sleep. This will be a 2 night sleep study (Night A will be without splint and Night B will be with splint). Therefore, the patient will sleep with the mouth guard one night and the monitoring device two nights. Subjects will also undergo CBCT airway imaging with and without splint.
  Arms: Modified farrar splint

SUMMARY:
The purpose of this study is to investigate the effects of mandibular occlusal stabilization splint (OSS) and modified farrar splint on sleep bruxism and respiratory indices and the effects of occlusal splints on the airway volume through imaging.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with sleep bruxism
* prescribed an occlusal splint

Exclusion Criteria:

* Less than 18 years old
* Secondary obstructive sleep apnea diagnosis
* Genetic disease that contributes to possible secondary obstructive sleep apnea
* Patient refuses to sign informed consent document
* Patient does not speak or read English
* More than two missing posterior teeth (excluding third molars)
* Presence of gross malocclusion

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-07-01 (Estimated); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in peripheral capillary oxygen saturation (SpO2) as measured by the MediByte device | Baseline(without device),with device
Change in pulse as measured by the MediByte device | Baseline(without device),with device
Change in airflow as measured by the MediByte device | Baseline(without device),with device
Change in chest plethysmography as measured by the MediByte device | Baseline(without device),with device
Change in abdomen plethysmography as measured by the MediByte device | Baseline(without device),with device
Change in masticatory muscle activity as measured by the MediByte device | Baseline(without device),with device

SECONDARY OUTCOMES:
Change in airway anatomy as measured by CBCT | Baseline(without device),with device

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Glick, DDS, Principal Investigator — The University of Texas Health Science Center, Houston

IPD SHARING:
Plan to Share IPD: No